CLINICAL TRIAL: NCT00348920
Title: The Effects of High Spinal Anesthesia on Hemodynamics, Stress Response, Renal Function and Post-operative Pain Control in Patients Undergoing Aortic Valve Replacement for Aortic Stenosis
Brief Title: The Effects of High Spinal Anesthesia on Heart Function, Stress Response and Pain Control in Aortic Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: St. Boniface Hospital (Other); Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Principal Investigator, Trevor William R. Lee, Site Leader, Dept. of Anesth, St. Boniface Hospital, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOTSA1
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Aortic Stenosis
Keywords: Aortic Valve; Aortic Stenosis; High Spinal Anesthesia; Total Spinal Anesthesia; Stress Response; Inflammatory Mediators; Renal Function; Hemodynamic Stability
MeSH Terms: conditions — Aortic Valve Stenosis; Fractures, Stress | interventions — Anesthesia, General; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- General Anesthesia (No Intervention): General Anesthesia includes administration of a routine cardiac anesthetic as per institutional norms.
- 2- High Spinal and General Anesthesia (Experimental): High Spinal and General Anesthesia includes a high dose intrathecal anesthetic administered prior to the induction of a standardized cardiac general anesthetic.
  Interventions: Procedure: High Spinal and General Anesthesia

INTERVENTIONS:
Procedure: High Spinal and General Anesthesia — Spinal bupivacaine 0.75% in dextrose, 6 mls (45mg) and preservative free morphine 3 mcg/kg (to a maximum of 300 mcg).
  Other Names: Bupivacaine; Epimorph
  Arms: 2- High Spinal and General Anesthesia

SUMMARY:
This study is looking at the effects of high spinal anesthesia (also known as total spinal anesthesia) combined with general anesthesia versus general anesthesia alone on the following:

Stress response: Patients undergoing aortic valve replacement surgery have a large incision and a complex operation where they must be placed on the heart-lung machine. The body reacts to the heart-lung machine, increasing the stress response.

High spinal anesthesia using local anesthetics when combined with general anesthesia has been shown to block some of the stress response to surgery and the response to the heart-lung machine. This study will examine if blood levels of stress hormones and also inflammatory mediators can be lowered with the use of high spinal anesthesia.

Heart function: High spinal anesthesia in combination with general anesthesia may help the heart work better when there is a narrowed valve (aortic stenosis). The heart may also have improved ability to pump blood with this anesthetic technique.

Lung function and post-operative pain control: After surgery, patients often have pain which prevents them from taking deep breaths and coughing. This can lead to pneumonia. This study will also examine if the post-operative pain relief provided by spinal morphine (given together with the spinal anesthetic) can provide any better pain control following surgery. By doing this, we want to see if patients can take bigger breaths after their surgery when spinal morphine is used, and try to prevent the complications that occur if patients are not able to breath deeply after surgery.

DETAILED DESCRIPTION:
It is hypothesized that high spinal anesthesia combined with general anesthesia decreases the intraoperative stress and inflammatory response and improve post-operative pain control and respiratory function in this patient population. It is also hypothesized that the technique will provide stable intraoperative hemodynamics during aortic valve replacement surgery.

Stress response: Levels of hormones such as epinephrine, norepinephrine and cortisol are elevated during cardiac surgery and on the initiation of cardiopulmonary bypass. This stress response has previously been shown to be blunted with the use of high spinal anesthesia when combined with general anesthesia in coronary artery bypass surgery patients (Lee, Grocott, et al).

Inflammatory response: In addition to the stress response there is also an accentuated inflammatory response. With contact of the patient's blood to the artificial bypass circuit, there is activation of various plasma protease pathways that generate multiple proinflammatory mediators. Complement levels and cytokine levels also rise. Clinical organ dysfunction involving the cardiovascular, pulmonary, renal and neurological systems can ultimately result. The effects of high spinal anesthesia on the inflammatory response that occurs with bypass have not been studied.

Hemodynamics: It has previously been shown that high-spinal anesthesia for coronary artery bypass surgery provides stable intra-operative hemodynamics (Kowalewski, MacAdams, et al; Lee, Grocott, et al.). Although the use of spinal anesthesia in patients with aortic stenosis has been considered to be relatively contra-indicated, total spinal anesthesia may actually improve cardiac function by decreasing systemic afterload and increasing myocardial contractility.

Post-operative analgesia and pulmonary function: The spinal administration of opioids, such as morphine, has been shown to improve post-operative pain management in patients having both cardiac and non-cardiac surgery (Jacobsohn, Lee, et al). Total spinal anesthesia with bupivacaine and spinal morphine combined with general anesthesia may also improve post-operative pain management and facilitate improved post-operative lung function.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery for aortic valve replacement due to aortic stenosis with or without CABG.

Exclusion Criteria:

* INR > 1.4, PTT > 40 seconds
* platelet count < 80, 000 per microlitre
* local infection or deformity at the site of administration of the spinal anesthetic
* raised intracranial pressure or evolving neurological deficit at the time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Stress response as measured by levels of circulating epinephrine, norepinephrine, and cortisol. | Multiple time points
Inflammatory response as measured by levels of circulating inflammatory mediators (e.g. interleukin-6, interleukin-8, interleukin-10, C-reactive protein, TNF-alpha). | Multiple time points
Blood glucose control (amount of insulin required to keep blood glucose 5-8 mmol/L). Renal function as measured by serum creatinine. | Multiple time points

SECONDARY OUTCOMES:
Vasopressor requirements to keep mean blood pressure between 60-80 mm Hg. | Multiple time points
Left ventricular wall motion score index as measured by TTE and TEE. | Multiple time points
Hemodynamics including cardiac output and cardiac index, heart rate, systemic arterial and pulmonary arterial blood pressures, central venous pressure, and systemic and pulmonary vascular resistance. | Multiple time points
Time to extubation. | Time of extubation

CONTACTS AND LOCATIONS:
Overall Officials: Trevor WR Lee, MD, Principal Investigator — Department of Anesthesia and Perioperative Medicine, St. Boniface General Hospital, University of Manitoba; Stephen E Kowalski, MD, Principal Investigator — Department of Anesthesia, Health Sciences Centre, University of Manitoba
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Lee TW, Grocott HP, Schwinn D, Jacobsohn E; Winnipeg High-Spinal Anesthesia Group. High spinal anesthesia for cardiac surgery: effects on beta-adrenergic receptor function, stress response, and hemodynamics. Anesthesiology. 2003 Feb;98(2):499-510. doi: 10.1097/00000542-200302000-00032. PMID 12552211
- [Background] Kowalewski R, MacAdams C, Froelich J, Neil S, Maitland A. Anesthesia supplemented with subarachnoid bupivacaine and morphine for coronary artery bypass surgery in a child with Kawasaki disease. J Cardiothorac Vasc Anesth. 1996 Feb;10(2):243-6. doi: 10.1016/s1053-0770(96)80246-1. No abstract available. PMID 8850406
- [Background] Jacobsohn E, Lee TW, Amadeo RJ, Syslak PH, Debrouwere RG, Bell D, Klock PA, Tymkew H, Avidan M; University of Manitoba Health Sciences Centre Cardiac Anesthesia Group. Low-dose intrathecal morphine does not delay early extubation after cardiac surgery. Can J Anaesth. 2005 Oct;52(8):848-57. doi: 10.1007/BF03021781. PMID 16189338
- [Derived] Lee TW, Kowalski S, Falk K, Maguire D, Freed DH, HayGlass KT. High Spinal Anesthesia Enhances Anti-Inflammatory Responses in Patients Undergoing Coronary Artery Bypass Graft Surgery and Aortic Valve Replacement: Randomized Pilot Study. PLoS One. 2016 Mar 1;11(3):e0149942. doi: 10.1371/journal.pone.0149942. eCollection 2016. PMID 26930568